CLINICAL TRIAL: NCT01081496
Title: Epidemiological Study to Evaluate the Prevalence of EGFR Mutation Status in Patients With Newly Diagnosed Locally Advanced or Metastatic NSCLC (Stage IIIB/IV Non-small Cell Lung Cancer)
Brief Title: Epidemiological Study to Evaluate the Prevalence of Epidermal Growth Factor Receptor (EGFR) Mutation Status in Patients With Newly Diagnosed Locally Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC)
Acronym: Spanish REASON
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-OES-DUM-2009/1
Record Dates: First submitted 2010-03-01; First posted 2010-03-05 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR mutation, Non-small cell lung carcinoma, Spain; Evaluate the prevalence of EGFR mutation status in patients with newly diagnosed locally advanced or metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To estimate the prevalence of EGFR mutation in a representative sample of patients with newly diagnosed stage IIIB/IV NSCLC in Spain (predominantly Caucasian ethnicity).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically confirmed locally advanced or metastatic NSCLC (stage IIIB/IV)

Exclusion Criteria:

* Mixed histology of small cell and non-small cell lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be recruited by Oncologist
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To estimate the prevalence of EGFR mutation in a representative sample of patients with newly diagnosed stage IIIB/IV NSCLC in Spain (predominantly Caucasian ethnicity).

SECONDARY OUTCOMES:
Correlate EGFR mutation status with clinico-pathological characteristics. The study will aim to determine the prevalence of EGFR M+ lung cancers in patients with clinico-pathological characteristics not commonly associated with EGFR mutation positivity
To describe different EGFR mutation methods used in Spain and testing turn around time associated
To determine the % of confirmed stage IIIB/IV NSCLC patients who cannot be tested for EGFR mutation and the reasons for not testing (% of EGFR Mnt)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gonzalez Arenas, Study Director — Medical Department. Mediclin-AstraZeneca. Spain
Locations (24):
- Spain (24):
  - Research Site, Santiago de Compostela, A Coruna
  - Research Site, Albacete, Albacete
  - Research Site, Alicante, Alicante
  - Research Site, Elche, Alicante
  - Research Site, Barcelona, Barcelona
  - Research Site, Cáceres, Caceres
  - Research Site, Santander, Cantabria
  - Research Site, Córdoba, Cordoba
  - Research Site, Girona, Girona
  - Research Site, Granada, Granada
  - Research Site, Jaén, Jaen
  - Research Site, Lugo, Lugo
  - Research Site, Madrid, Madrid
  - Research Site, Málaga, Malaga
  - Research Site, Murcia, Murcia
  - Research Site, Pamplona, Navarre
  - Research Site, Pontevedra, Pontevedra
  - Research Site, Vigo, Pontevedra
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Salamanca, Salamanca
  - Research Site, Seville, Sevilla
  - Research Site, Reus, Tarragona
  - Research Site, Valencia, Valencia
  - Research Site, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Esteban E, Majem M, Martinez Aguillo M, Martinez Banaclocha N, Domine M, Gomez Aldaravi L, Juan O, Cajal R, Gonzalez Arenas MC, Provencio M. Prevalence of EGFR mutations in newly diagnosed locally advanced or metastatic non-small cell lung cancer Spanish patients and its association with histological subtypes and clinical features: The Spanish REASON study. Cancer Epidemiol. 2015 Jun;39(3):291-7. doi: 10.1016/j.canep.2015.02.003. Epub 2015 Mar 9. PMID 25766256